CLINICAL TRIAL: NCT04989439
Title: Comparison of Computertomography Scan, Electrical Impedance Tomography, and Ultrasound of the Lung in Infants - a Prospective Explorative Observational Study
Brief Title: Comparison of Computertomography Scan, Electrical Impedance Tomography, and Ultrasound of the Lung in Infants
Status: Recruiting | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Tobias Werther, Principal Investigator, Medical University of Vienna
Other Study IDs: 1565/2021
Record Dates: First submitted 2021-07-25; First posted 2021-08-04 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Infant ALL; Computed Tomography; Electric Impedance; Ultrasonography; Lung Injury
Keywords: CT, electrical impedance tomography, ultrasound
MeSH Terms: conditions — Lung Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Electrical impedance tomography and ultrasonography of the lung — Both EIT and LUS are non-invasive methods and do not pose any additional risk for the patient. The LuMon System with pediatric EIT belts (LuMon Belt, Sentec, Landquart, Switzerland) will be used. The belt will be placed on the thorax circumference of the infant and connected to the LuMonConnector (Sentec, Landquart, Switzerland). Small electrical currents (3 mA, 198 kHz) will be repetitively injected in rotation through adjacent electrode pairs, and voltage changes will be measured by all passive electrodes pairs (scan rate 48 Hz). Changes in lung electrical impedance will be continuously recorded for 5 minutes. EIT data will be analyzed off-line using Matlab (Mathworks, Natick, Massachusetts, USA). The regional tidal volume distribution, the homogeneity of tidal ventilation distribution, regional respiratory system compliance, and alveolar overdistension and collapse will be assessed. LUS will be performed by experienced users, with a 10 MHz linear transducer.

SUMMARY:
The study focuses on regional lung examination, in particular on the differentiation between collapsed and hyperinflated lung areas. The purpose of the study is to elaborate common and discriminative elements between different lung imaging modalities in infants and to generate hypotheses for the bedside use of EIT and LUS in infants.

DETAILED DESCRIPTION:
Lung imaging has become increasingly important across medical specialties for diagnostic, monitoring, and investigative purposes in acute respiratory distress syndrome (ARDS). Lung computer tomography (CT) is the gold standard chest imaging technique to evaluate lung morphology and to perform a quantitative analysis of lung tissue aeration and recruitment. In the last decades, electrical impedance tomography (EIT) has gained a lot of attention in monitoring functional lung parameters. EIT is a non-invasive, bedside radiation-free functional imaging modality for continuous monitoring of lung ventilation and perfusion. Functional chest examinations with EIT are considered clinically relevant, especially for monitoring regional lung ventilation in patients with respiratory support, but also to assess aeration in preterm and term infants. In comparison with dynamic CT, EIT proved to be useful in bedside adjustments of mechanical ventilation with immediate feedback in adult patients. EIT lacks the spatial resolution of other imaging modalities but it is compact in size, uses no ionizing radiation, and gives functional images with high temporal resolution. As CT scans expose patients to ionizing radiation, there are no investigative studies comparing EIT with CT scans in newborns and infants. This would be useful, particularly, for correlating the reference impedance image with a CT scan to correctly calibrate anatomical structures and to differentiate between dependent and non-dependent lung areas. Likewise, lung ultrasound (LUS) has been increasingly used for the diagnosis of different lung conditions. Some validation studies compared LUS with CT scans and classified LUS to be a valid tool to assess regional and global lung aeration also in newborns. To our knowledge, there are no comparative studies between EIT and LUS in newborns and infants.

The main objective is to compare different lung imaging modalities in infants with and without lung disease using the CT scan as reference method. The study focuses on regional lung examination. The purpose of the study is to elaborate common and discriminative elements between different lung imaging modalities in infants and to generate hypotheses for the bedside use of EIT and LUS in this group of patients.

The CT scan is part of the routine care of the participants. No additional CT examinations will be performed for this study. LUS and EIT will be performed immediately before or after the planned CT scan. Both LUS and EIT measurements will be performed with mobile devices and will take approximately 20 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized at the Department of Pediatrics of the Medical University of Vienna who will get a CT scan of the thorax.
* Patients aged up to 12 months

Exclusion Criteria:

* Unstable cardiovascular, respiratory and/or neurological conditions.
* Sternotomy during the previous 15 days.
* Thoracic skin lesions or wounds (including burns) on the thorax, where the EIT-electrode-belt would be placed.

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants receiving a CT scan of the thorax.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2021-07-19 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparison between CT and EIT | through study completion, an average of 1 year
  Estimate difference of lung cross-section between CT scan and EIT
Comparison between CT and LUS | through study completion, an average of 1 year
  Comparison of diagnosis (presence of pathologic patterns including pneumothorax, emphysema, atelectasis, consolidation, ground glass opacity, bronchial wall thickening and/or dilatation) in CT and LUS

SECONDARY OUTCOMES:
Comparison between EIT and LUS | through study completion, an average of 1 year
  Comparison of dynamic parameters of dorsal and ventral regions

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Werther, MD, PhD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pesenti A, Musch G, Lichtenstein D, Mojoli F, Amato MBP, Cinnella G, Gattinoni L, Quintel M. Imaging in acute respiratory distress syndrome. Intensive Care Med. 2016 May;42(5):686-698. doi: 10.1007/s00134-016-4328-1. Epub 2016 Mar 31. PMID 27033882
- [Background] Ball L, Vercesi V, Costantino F, Chandrapatham K, Pelosi P. Lung imaging: how to get better look inside the lung. Ann Transl Med. 2017 Jul;5(14):294. doi: 10.21037/atm.2017.07.20. PMID 28828369
- [Background] Caironi P, Gattinoni L. How to monitor lung recruitment in patients with acute lung injury. Curr Opin Crit Care. 2007 Jun;13(3):338-43. doi: 10.1097/MCC.0b013e32814db80c. PMID 17468568
- [Background] Chiumello D, Mongodi S, Algieri I, Vergani GL, Orlando A, Via G, Crimella F, Cressoni M, Mojoli F. Assessment of Lung Aeration and Recruitment by CT Scan and Ultrasound in Acute Respiratory Distress Syndrome Patients. Crit Care Med. 2018 Nov;46(11):1761-1768. doi: 10.1097/CCM.0000000000003340. PMID 30048331
- [Background] Frerichs I, Weiler N. Electrical impedance tomography: the next game level*. Crit Care Med. 2012 Mar;40(3):1015-6. doi: 10.1097/CCM.0b013e31823d7849. No abstract available. PMID 22343863
- [Background] Frerichs I, Amato MB, van Kaam AH, Tingay DG, Zhao Z, Grychtol B, Bodenstein M, Gagnon H, Bohm SH, Teschner E, Stenqvist O, Mauri T, Torsani V, Camporota L, Schibler A, Wolf GK, Gommers D, Leonhardt S, Adler A; TREND study group. Chest electrical impedance tomography examination, data analysis, terminology, clinical use and recommendations: consensus statement of the TRanslational EIT developmeNt stuDy group. Thorax. 2017 Jan;72(1):83-93. doi: 10.1136/thoraxjnl-2016-208357. Epub 2016 Sep 5. PMID 27596161
- [Background] Victorino JA, Borges JB, Okamoto VN, Matos GF, Tucci MR, Caramez MP, Tanaka H, Sipmann FS, Santos DC, Barbas CS, Carvalho CR, Amato MB. Imbalances in regional lung ventilation: a validation study on electrical impedance tomography. Am J Respir Crit Care Med. 2004 Apr 1;169(7):791-800. doi: 10.1164/rccm.200301-133OC. Epub 2003 Dec 23. PMID 14693669
- [Background] Wolf GK, Gomez-Laberge C, Rettig JS, Vargas SO, Smallwood CD, Prabhu SP, Vitali SH, Zurakowski D, Arnold JH. Mechanical ventilation guided by electrical impedance tomography in experimental acute lung injury. Crit Care Med. 2013 May;41(5):1296-304. doi: 10.1097/CCM.0b013e3182771516. PMID 23474677
- [Background] Muders T, Luepschen H, Zinserling J, Greschus S, Fimmers R, Guenther U, Buchwald M, Grigutsch D, Leonhardt S, Putensen C, Wrigge H. Tidal recruitment assessed by electrical impedance tomography and computed tomography in a porcine model of lung injury*. Crit Care Med. 2012 Mar;40(3):903-11. doi: 10.1097/CCM.0b013e318236f452. PMID 22202705
- [Background] Raimondi F, Yousef N, Migliaro F, Capasso L, De Luca D. Point-of-care lung ultrasound in neonatology: classification into descriptive and functional applications. Pediatr Res. 2021 Sep;90(3):524-531. doi: 10.1038/s41390-018-0114-9. Epub 2018 Jul 20. PMID 30127522
- [Background] Liu J, Chen SW, Liu F, Li QP, Kong XY, Feng ZC. The diagnosis of neonatal pulmonary atelectasis using lung ultrasonography. Chest. 2015 Apr;147(4):1013-1019. doi: 10.1378/chest.14-1306. PMID 25341049
- [Background] Zieleskiewicz L, Markarian T, Lopez A, Taguet C, Mohammedi N, Boucekine M, Baumstarck K, Besch G, Mathon G, Duclos G, Bouvet L, Michelet P, Allaouchiche B, Chaumoitre K, Di Bisceglie M, Leone M; AZUREA Network. Comparative study of lung ultrasound and chest computed tomography scan in the assessment of severity of confirmed COVID-19 pneumonia. Intensive Care Med. 2020 Sep;46(9):1707-1713. doi: 10.1007/s00134-020-06186-0. Epub 2020 Jul 29. PMID 32728966
- [Background] Sophocleous L, Frerichs I, Miedema M, Kallio M, Papadouri T, Karaoli C, Becher T, Tingay DG, van Kaam AH, Bayford R, Waldmann AD. Clinical performance of a novel textile interface for neonatal chest electrical impedance tomography. Physiol Meas. 2018 Apr 26;39(4):044004. doi: 10.1088/1361-6579/aab513. PMID 29516865
- [Background] Adler A, Arnold JH, Bayford R, Borsic A, Brown B, Dixon P, Faes TJ, Frerichs I, Gagnon H, Garber Y, Grychtol B, Hahn G, Lionheart WR, Malik A, Patterson RP, Stocks J, Tizzard A, Weiler N, Wolf GK. GREIT: a unified approach to 2D linear EIT reconstruction of lung images. Physiol Meas. 2009 Jun;30(6):S35-55. doi: 10.1088/0967-3334/30/6/S03. Epub 2009 Jun 2. PMID 19491438
- [Background] Brat R, Yousef N, Klifa R, Reynaud S, Shankar Aguilera S, De Luca D. Lung Ultrasonography Score to Evaluate Oxygenation and Surfactant Need in Neonates Treated With Continuous Positive Airway Pressure. JAMA Pediatr. 2015 Aug;169(8):e151797. doi: 10.1001/jamapediatrics.2015.1797. Epub 2015 Aug 3. PMID 26237465